CLINICAL TRIAL: NCT02002936
Title: Phase I Clinical Trial of SyB C-1101 in Patients With Myelodysplastic Syndrome - Extension Study
Brief Title: Long Term Safety Study of SyB C-1101 in Patients With Recurrent/Relapsed or Refractory Myelodysplastic Syndrome (MDS) - Extension Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SymBio Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012004
Record Dates: First submitted 2013-12-01; First posted 2013-12-06 (Estimated); Results first posted 2016-12-12 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-01

CONDITIONS: Myelodysplastic Syndrome
MeSH Terms: conditions — Myelodysplastic Syndromes

ARMS (1):
- SyB C-1101 (Experimental)
  Interventions: Drug: SyB C-1101

INTERVENTIONS:
Drug: SyB C-1101 — SyB C-1101（rigosertib sodium） will be administered orally twice daily for 14 consecutive days, followed by 7-day observation period. The treatment period of 21 days (14 days of administration + 7 days of observation) constitutes 1 cycle.
  The dose at cycle 6 in the study 2012002 will be the dose (if needed, the dose can be reduced) at the first cycle in this study (cycle 7).
  From cycle 8 on, the dose of SyB C-1101 will be reduced, delayed, or discontinued according to adverse events and results of observation at the previous cycle.

SUMMARY:
This is an extension study to investigate long term safety and efficacy of SyB C-1101 when orally administered every 3 weeks, twice daily for 14 consecutive days to the patients who have completed 6 cycles in the study 2012002 whose purpose is to investigate tolerability of SyB C-1101 when administered orally in patients with recurrent/relapsed or refractory myelodysplastic syndrome.

ELIGIBILITY:
Inclusion Criteria:

Patients must satisfy the following conditions listed below.

1. Patients enrolled in the study 2012002 of SyB C-1101 in Patients With Myelodysplastic Syndrome.
2. Patients who were not judged as disease progression* nor progressive disease/relapse** at the end of the cycle 6 in the study 2012002. * hematologic remission according to IWG 2006 criteria ** hematologic improvement according to IWG 2006 criteria
3. Patients who met the continuation criteria*** after Cycle 6 week 3 (Day 22±3) in the study 2012002.

   ***defined in the study 2012002 protocol "4.5 Criteria for Transition to the Next Cycle "
4. Patients who can be expected to survive at least three months or longer.
5. Patients who have score of 0 to 2 in Eastern Cooperative Oncology Group (ECOG) Performance Status (PS).
6. Patients with adequate function in major organs (heart, lungs, liver, kidneys, etc.).

   * Aspartate aminotransferase (AST): no more than 3.0 times the upper boundary of the reference range at each institution
   * Alanine aminotransferase (ALT): no more than 3.0 times the upper boundary of the reference range at each institution
   * Total bilirubin: no more than 1.5 times the upper boundary of the reference range at each institution
   * Serum creatinine: no more than 1.5 times the upper boundary of the reference range at each institution
   * ECG: no abnormal findings requiring treatment
   * Echocardiography: no abnormal findings requiring treatment
7. Patients who personally signed an informed consent document for participation in this study.

Exclusion Criteria:

Patients who satisfy any of the following conditions after Cycle 6 week 3 (Day 22±3) in the study 2012002 will not be enrolled in the study.

1. Patients with anemia caused by factors other than MDS(hemolytic anemia, gastrointestinal hemorrhage, etc.).
2. Patients with obvious infectious diseases (including viral infections).
3. Patients with serious complications (liver failure, renal failure, etc.).
4. Patients with a complication of serious heart disease (myocardial infarction, ischemic heart disease, etc.)
5. Patients with a serious gastrointestinal condition (severe or significant nausea/vomiting, diarrhea, etc.)
6. Patients with serious bleeding tendencies (disseminated intravascular coagulation (DIC), internal hemorrhage, etc.).
7. Ascites or pleural fluid requiring active medical management including paracentesis, or hyponatremia (defined as serum sodium value of < 130 mEq/L).
8. Patients with known allergy to polyethylene glycol or gelatin capsules.
9. Patients with an addiction to a legal or illegal drug, or with alcohol dependency.
10. Patients who are nursing, pregnant or may become pregnant, or lactating mothers.
11. Patients who have not consented to the following contraceptive measures. Patients will avoid sexual intercourse with sexual partners or should use the following contraceptive methods in these time periods: for male patients during the administration period of the trial and for six months after the end of administration; female patients during the administration period of the trial and until a second menstrual period is confirmed after the end of administration (or in the case of female patients with no menstrual period, for two months after the end of administration). 1) Male patients: Patients will always use a condom.

    For effective contraception, it is recommended that the female partner also use the contraceptive methods for female patients. 2) Female patients: Female patients who may become pregnant should use one or more types of the following contraceptive methods. In addition, the male partner will always use a condom.
    * Oral contraceptive (birth control pills)
    * Intrauterine device (IUD)
    * Tubal ligation
12. Other patients judged to be unsuitable by an investigator or sub-investigators.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2013-08; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katsuhisa Goto, Study Director — SymBio Pharmaceuticals
Locations (4):
- Japan (4):
  - Research Site, Nagoya, Aichi-ken
  - Research Site, Isehara, Kanagawa
  - Research Site, Kyoto, Kyoto
  - Research Site, Sendai, Miyagi

RESULTS

PARTICIPANT FLOW:
Groups:
- SyB C-1101: SyB C-1101 （rigosertib sodium）:
  Following Cycle 6 of Study 2012002, the treatment in this study was initiated. One cycle was defined as a 21-day cycle; 14-day oral administration of SyB C-1101 twice daily (Days 1 to 14) followed by a 1-week observation period (Days 15 to 21). The starting dose of SyB C-1101 in this study (Cycle 7) was the same as that was determined for the next cycle in Cycle 6 of Study 2012002.
Period: Overall Study
Arm/Group | SyB C-1101
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | SyB C-1101
Number analyzed (Participants) | 1
Age, Customized [Number; unit: participants]
  50-59 years | 1
  60-69 years | 0
  70-79 years | 0
  80-years | 0
Gender [Count of Participants; unit: Participants]
  Female | 0
  Male | 1

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events
Description: Total number affected by any adverse events (details are presented in adverse event section)
Time Frame: Up to 3 years
Measure: Number; unit: participants
Arm/Group | SyB C-1101
Number analyzed (Participants) | 1
participants | 1

2. Secondary Outcome: Total Efficacy in Hematologic Remission (IWG2006 Criteria)
Description: SD (stable disease): according to International Working Group 2006 response criteria for myelodysplastic syndrome, SD was defined as a failure to achieve "complete remission" or "partial remission," but no evidence of progression for > 8 weeks.
Time Frame: Up to 3 years
Measure: Number; unit: participants
Arm/Group | SyB C-1101
Number analyzed (Participants) | 1
participants | 1

3. Secondary Outcome: Total Efficacy in Hematologic Improvement Ratio According to IWG 2006 Criteria.
Description: NCA (not considered assessable): no evidence of HI-E (hematologic improvement-erythroid), HI-P (hematologic improvement-platelet), HI-N (hematologic improvement-neutorophil), progressive disease, or relapse.
Time Frame: Up to 3 years
Measure: Number; unit: participants
Arm/Group | SyB C-1101
Number analyzed (Participants) | 1
participants | 1

4. Secondary Outcome: Cytogenetic Response Ratio According to IWG 2006 Criteria
Description: NCA (not considered assessable): no cytogenetic response
Time Frame: Up to 3 years
Measure: Number; unit: participants
Arm/Group | SyB C-1101
Number analyzed (Participants) | 1
participants | 1

5. Secondary Outcome: Overall Survival
Description: Survived
Time Frame: Up to 3 years
Measure: Number; unit: participants
Arm/Group | SyB C-1101
Number analyzed (Participants) | 1
participants | 1

6. Secondary Outcome: Changes in Clinical Laboratory Test Results
Description: Clinically significant changes
Time Frame: Up to 3 years
Measure: Number; unit: participants
Arm/Group | SyB C-1101
Number analyzed (Participants) | 1
participants | 0

ADVERSE EVENTS:
Arm/Group | SyB C-1101
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SyB C-1101 (N=1)
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Asthenopia (Eye disorders) | 1 (1)
Ligament sprain (Musculoskeletal and connective tissue disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Periodontitis (Injury, poisoning and procedural complications) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No